CLINICAL TRIAL: NCT03971292
Title: Interest of High-throughput Sequencing of RNAs for the Diagnosis of Heterogeneous Genetic Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7004
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: DNA Sequencing; Diagnosis of Genetic Diseases of Heterogeneous Origin
MeSH Terms: interventions — Sequence Analysis, RNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Validation phase: The project will proceed in two phases: a validation test phase including 5 patients of known genotype and a prospective phase including 10 patients.
  Interventions: Genetic: RNA sequencing
- Prospective phase: The project will proceed in two phases: a validation test phase including 5 patients of known genotype and a prospective phase including 10 patients.
  Interventions: Genetic: RNA sequencing

INTERVENTIONS:
Genetic: RNA sequencing — Testing interest of messenger RNA sequencing for the etiological diagnosis of unresolved patients after sequencing coding regions.

SUMMARY:
The advent of high throughput genomic DNA sequencing has led to major advances in the diagnosis of genetic diseases of heterogeneous origin. Thus, our hospital laboratory has developed in recent years several diagnostic tests based on the targeted sequencing of coding sequences of gene panels (from about twenty genes for DNA repair diseases to nearly five hundred genes for the intellectual disability). These targeted analyzes, carried out by capture, have thus solved 25 to 80% of the cases according to the indications, without allowing the diagnosis of the totality of the patients.

For these negative cases, the search for mutations in the coding sequences was then extended to Whole Exome Sequencing, thus providing several additional diagnoses.

Patients still remain without diagnosis after this exome study. These could be complex cases of genetic or even non-genetic origin, but also monogenic pathologies linked to mutations that are not identifiable by coding sequence analyzes, and especially affecting messenger RNAs.

ELIGIBILITY:
Inclusion criteria common to all participants:

* Patient minor or major
* Patient suffering from a pathology studied in the laboratory by high throughput sequencing: intellectual disability, myopathies, neurosensory disease (Bardet-Biedl syndrome, retinitis pigmentosa, ....), DNA repair diseases (Cockayne syndrome, ...)
* Sampling allowing the extraction of available RNA (or RNA available in the bank)
* Patient (or its legal representative) having already given their consent, on the one hand for carrying out genetic analyzes to determine the cause of their disease, and on the other hand for the conservation of part of their non used for further use in order to continue diagnostic investigations in the light of evolving knowledge and for research purposes.
* Patient (or its legal representative) agreeing to use data from his medical file and those associated with genetic diagnosis for research purposes
* Patient affiliated to a social security scheme Inclusion criteria for the test phase
* Pertogenous mutation (s) known Inclusion criteria for the prospective phase
* Magnetic molecular diagnosis, after the usual investigations (high-throughput sequencing of a panel of genes on genomic DNA, sequencing of exome, or even genome.

Non-inclusion criteria:

◾ Refusal of the patient (or his / her legal representative) to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient suffering from a pathology studied in the laboratory by high throughput sequencing: intellectual disability, myopathies, neurosensory disease (Bardet-Biedl syndrome, retinitis pigmentosa, ....), DNA repair diseases (Cockayne syndrome, ...)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
RNA sequencing | 3 years
  testing interest of messenger RNA sequencing for the etiological diagnosis of unresolved patients after sequencing of coding regions, and its integration into hospital routine in order to improve the diagnosis of heterogeneous genetic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided